CLINICAL TRIAL: NCT00812760
Title: Effect of Levodopa on Human Multifocal Electroretinogram
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Michael Wolzt, Department of Clinical Pharmacology, Medical University of Vienna
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OPHT-220501
Record Dates: First submitted 2008-12-18; First posted 2008-12-22 (Estimated); Last update posted 2008-12-22 (Estimated); Status verified 2008-12

CONDITIONS: Retinal Diseases
Keywords: Electroretinography; levodopa
MeSH Terms: conditions — Retinal Diseases | interventions — Levodopa; benserazide, levodopa drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: levodopa

INTERVENTIONS:
Drug: levodopa — 1 tablet of 200 mg levodopa plus 50 mg benserazide
  Other Names: Madopar

SUMMARY:
It is known that dopamine is a functional neuromodulator at several levels of the visual system. Dopamine seems to be involved in the organization of the ganglion cell and the bipolar cell receptive fields and modulation of physiological activity of photoreceptors. There is evidence for the functional significance of dopaminergic modulation of visual sensitivity in humans which confirms the hypothesis that dopamine plays an important role in retinal light adaptation as well as in motion and contrast sensitivity function. The electrophysiological effects of dopamine, various dopamine antagonist and levodopa in animals and humans have been investigated by means of visual evoked potentials and electroretinograms. The multifocal ERG technique, developed by Sutter et al. allows a rapid, simultaneous recording of focal ERGs from multiple retinal locations. Although this technique is relatively new, it has already provided insights into the mechanisms of retinal diseases (e.g. involvement of visual system in Parkinson disease), but until now there is no data on influence of dopaminergic substances on mERG.

ELIGIBILITY:
Inclusion Criteria:

* Men aged between 19 and 35 years, nonsmokers
* Body mass index between 15th and 85th percentile
* Normal findings in the medical history and physical examination unless the investigator considers an abnormality to be clinically irrelevant
* Normal laboratory values unless the investigator considers an abnormality to be clinically irrelevant
* Normal ophthalmic findings, ametropia < 3 Dpt

Exclusion Criteria:

* Regular use of medication, abuse of alcoholic beverages, participation in a clinical trial in the 3 weeks preceding the study
* Treatment in the previous 3 weeks with any drug
* Symptoms of a clinically relevant illness in the 3 weeks before the first study day
* History of hypersensitivity to the trial drug or to drugs with a similar chemical structure
* History or presence of gastrointestinal, liver or kidney disease, or other conditions known to interfere with, distribution, metabolism or excretion of study drugs
* Blood donation during the previous 3 weeks

Ages: 19 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2001-10; Primary Completion 2003-10 (Actual); Study Completion 2003-10 (Actual)

PRIMARY OUTCOMES:
Retinal activity (mERG amplitude) | 5 measurements on both study days

SECONDARY OUTCOMES:
Retinal activity (mERG latency) | 5 measurements on both study days
Dopamine and levodopa plasma levels | on both study days

CONTACTS AND LOCATIONS:
Overall Officials: Michael Wolzt, MD, Principal Investigator — Department of Clinical Pharmacology, Medical University of Vienna
Locations (1):
- Department of Clinical Pharmacology, Medical University of Vienna, Vienna, Austria